CLINICAL TRIAL: NCT07277959
Title: Novel Use of Grommet Tube in the Treatment of Odontogenic Cysts Marsupialization
Brief Title: Marsupialization of Odontogenic Cysts
Status: Completed | Type: Observational
Sponsor: University Of Anbar (Other)
Responsible Party: Principal Investigator, Batool Abdulnasser Ismail, Postgraduate Student, Department of Oral Surgery, University Of Anbar
Other Study IDs: Ref. 236, in 25-12-2024
Record Dates: First submitted 2025-11-28; First posted 2025-12-11 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-01

CONDITIONS: Odontogenic Cysts Marsupialization

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: novel use of Grommet tube — The intervention consisted of performing conventional marsupialization of the odontogenic cyst followed by the novel placement of a ventilation Grommet tube to maintain long-term patency of the surgical window. After administration of local anesthesia, a small bony window was created over the thinnest cortical area of the cyst to expose the cystic cavity. The cyst lining was incised then the tube was placed

SUMMARY:
To evaluate the efficacy of the Grommet tube by measuring the rate of reduction in cyst size, assess patients satisfaction, and evaluate the occurrence of complications.

ELIGIBILITY:
Inclusion Criteria:

* Pathological diagnosis of odontogenic cyst
* Indicated for marsupialization
* Patients aged from 15 to 60 years

Exclusion Criteria:

* Soft tissue cysts.
* Patients with systemic diseases affecting bone healing.
* Patients non-compliance with follow up visits.
* Patients with a history of neck and head radiotherapy or patients on chemotherapy.
* Patients taking antiresorptive drugs or corticosteroids.

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The group of patients in this study consisted of individuals diagnosed with odontogenic cysts who are indicated for marsupialization procedure. Ten patients were enrolled in this study.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2025-01-02 (Actual); Primary Completion 2025-10-10 (Actual); Study Completion 2025-10-20 (Actual)

PRIMARY OUTCOMES:
Reduction in Cyst Size | 6 months
  Cyst volume will be measured using CBCT and 3D Slicer segmentation at baseline and 6 months after marsupialization. Percentage reduction in cyst size will be calculated.
Patient Satisfaction | Time Frame: 6 months
  Patient satisfaction will be assessed using a validated questionnaire (e.g., 3-point Likert scale) at 6 months.
Occurrence of Complications | Time Frame: 6 months
  The presence of postoperative complications (infection, device displacement, or soft tissue overgrowth) will be recorded clinically at follow-up visits.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Anbar-college of dentistry, Ramadi, Iraq